CLINICAL TRIAL: NCT03407859
Title: Sequential Treatment With CD20/CD22/CD10-CART After CD19-CART Treatment Base on MRD in Relapsed/Refractory B-ALL
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2016-XYNK-002
Record Dates: First submitted 2017-04-09; First posted 2018-01-23 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Therapy Related Leukemia
Keywords: CD19-CART; CD20-CART; CD10-CART; CD22-CART; Relapsed/Refractory B-ALL; MRD; CD70-CART
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequential therapy with different CART (Experimental): Sequential therapy With different CART including one kind of CD20/CD22/CD10-CART After CD19-CART therapy in CD19-negative relapse ALL patients, subjects will receive 1-5 x 10^6/Kg transduced CAR T cells at one time.
  Interventions: Biological: Sequential Treatment With different CART

INTERVENTIONS:
Biological: Sequential Treatment With different CART — Sequential Treatment With CD20/CD22/CD10-CART After CD19-CART Treatment in Relapsed/Refractory B-ALL

SUMMARY:
CD19-negative B-ALL relapses after CD19 CAR T-cell treatment have occurred in some patients. CD20/CD22/CD10 is still expressed in CD19 negative B-ALL cells which means these CD molecules may become new targets in treatment of CD19-negative relapse of B-ALL. Thus sequential treatment with CD20/CD22/CD10-CART after CD19-CART treatment in relapsed/refractory B-ALL will kill and eliminate CD19 negative B-ALL cells and prolong the remission time.

DETAILED DESCRIPTION:
B-cell acute lymphoblastic leukemia is the most common type of leukemia and the prognosis of relapsed/refractory B-ALL is poor. Chimeric Antigen Receptor-transduced T cell (CAR-T) therapy is one of revolutionary targeted immunotherapy. CD19 CAR-T is the most commonly used engineered T cell in B-ALL. The treatment effect is significant and far more than traditional therapy in relapsed/refractory B-ALL. However, the remission time after CD19 CAR-T infusion is short.CD19-positive and CD19-negative B-ALL relapses after CD19 CAR T-cell treatment have occurred in some patients The cause of relapse after CAR-T infusion is minimal residual disease (MRD) which will induce CD19 negative relapse. CD20/CD22/CD10 is still expressed in CD19 negative B-ALL cells which means these CD molecules may become new targets in treatment of CD19 negative relapse of B-ALL. Thus sequential treatment with CD20/CD22/CD10-CART after CD19-CART treatment in relapsed/refractory B-ALL will kill and eliminate CD19 negative B-ALL cells and prolong the remission time.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/Refractory B-ALL patients
2. Did not achieve complete remission after 2 times of standard plan chemotherapy
3. Relapsed after first induction chemotherapy
4. Did not response to chemotherapy before HSCT or relapsed after HSCT
5. Cannot receive allo-HSCT or refuse to receive allo-HSCT
6. Cell phenotype is CD19 and CD20/CD22/CD10/CD70 positive (single or combined)
7. Estimated survival time is more than 3 months in leukemia
8. Volunteered for this clinical trail and signed a consent form

Exclusion Criteria:

1. MRD was negative while the cell phenotype was CD19 expressed
2. Patients with severe insufficient cardiac, pulmonary and hepatorenal functions
3. Patients with severe mental illness, neurological disease or infectious disease
4. Patients with GVHD was taking immunosuppressants
5. Pregnant or lactating women
6. Patients have received other genetic therapy products
7. Transfection efficiency was less than 30%
8. Any situation may do harm to the subjects or interfere the results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events that Are related to treatment | 2 years
  Determine the toxicity profile of the CD19-targeted and CD20/CD22/CD10-targeted CAR-T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Estimate 2 year overall survival(OS) after infusion of CD19-CART and sequential treatment | 2 years
  To estimate 2 year overall survival(OS) after CD19-CART infusion and sequential treatment with Relapsed/Refractory B-ALL
Estimate relapse rate after infusion of CD19-CART and sequential treatment | 4 years
  To estimate relapse rate after CD19-CART infusion and sequential treatment with Relapsed/Refractory B-ALL
Estimate 2 year progression free survival after infusion of CD19-CART and sequential treatment | 2 years
  To estimate 2 year progression free survival (PFS) after CD19-CART infusion and sequential treatment with Relapsed/Refractory B-ALL

CONTACTS AND LOCATIONS:
Overall Officials: Yanjie He, Ph.D, Principal Investigator — Zhujiang Hospital
Locations (1):
- Southern Medical University Zhujiang Hospital, Guangdong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No